CLINICAL TRIAL: NCT06216600
Title: Women Focused Encounters for Resilience Independence Strength and Eudaimonia
Acronym: WE RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Christie's Place (Other); By His Stripes Wellness Center (Other); Sister Love (Other); APLA Health (Unknown)
Responsible Party: Principal Investigator, Maile Young Karris, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 808061
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections; Substance Use; Trauma; Medication Adherence
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Wounds and Injuries; Medication Adherence | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Type 1 hybrid study randomizing particpants 1:1 to either WE RISE or control (list of resources). Followed by one arm observational study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study investigators and outcomes assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WE RISE Intervention (Experimental): Participants will undergo WE RISE intervention: twice a week for 8 week combination delivery of acceptance and commitment therapy + exercise + social suppot.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Body weight circuit training; Behavioral: Empathetic social support
- Control (Active Comparator): Participants will receive standard of care which would be referrals to local opportunites for therapy, exercise and social support.
  Interventions: Other: Control - list of resources
- Observational (Experimental): Observational study of participants undergoing WE RISE adapted for sustainability.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Body weight circuit training; Behavioral: Empathetic social support

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Participants will undergo ACT in combination with exercise and social support.
  Arms: Observational; WE RISE Intervention
Behavioral: Body weight circuit training — Participants will learn and undergo body weight circuit training in combination with ACT and social support.
  Arms: Observational; WE RISE Intervention
Behavioral: Empathetic social support — Study participants will participate in empathetic social support
  Arms: Observational; WE RISE Intervention
Other: Control - list of resources — A local list of resources to access exercise, therapy and social support will be provided.
  Arms: Control

SUMMARY:
The goal of this combination Type 1 hybrid and observational study is to evaluate the impact of a peer delivered intervention of acceptance and comittment therapy(ACT) + exercise + social support to address the substance (ab)use, violence, and AIDS/HIV (SAVA) to improve medication adherence for women living with HIV (WLWH). This intervention will be implemented by community based organizations that focus on WLWH across four counties. The main question it aims to answer are:

* Will peer provision of ACT, exercise, and social support improve medication adherence for WLWH?
* Will community based organizations be able to sustain the intervention after research is completed, and what changes will need to be made to sustain th eintervention.

DETAILED DESCRIPTION:
In the U.S. women living with HIV (WLWH) are less likely to engage in HIV care, be on antiretroviral therapy (ART), and achieve sustained viral suppression compared to men. The Substance (Ab)use, Violence/trauma, and HIV/AIDS (SAVA) syndemic is proposed to primarily contribute to gender-based differences in HIV outcomes.To meaningful address SAVA requires interventions that focus on each epidemic and transdiagnostic processes (shared mediators) including mood (depression/anxiety), HIV stigma, and loneliness. The Women focused Encounters for Resilience, Independence, Strength, and Eudaimonia (WE RISE) intervention addresses SAVA by employing peer navigator (PN) delivered group-based acceptance and commitment therapy (ACT) + exercise + empathetic social support.

The goal of this proposal is to evaluate and implement WE RISE for WLWH across four sites in Ending the HIV Epidemic (EHE) jurisdictions (San Diego, CA; Charlotte, NC; Atlanta, GA and Los Angeles, CA). This study is guided by a study advisory board (SAB) of 12 women living with and/or otherwise affected by HIV.

At each site peers will be trained at the University of California San Diego (UCSD) to provide ACT, exercise and social support thorugh didactic and experiential experiences and a workbook that guides them through the intervention. WE RISE delivery will be monitored by experts at UCSD and peers provided feedback through 6 months to encourage the devleopment of mastery.

The first phase of WE RISE is a type 1 hybrid study that will involve randomizing participants 1:1 to the WE RISE intervention or a local curated list of resources that focus on providing HIV care, therapy, exercise and social support. All participants in this phase will undergo assessments (HIV adherence, trauma symptoms, substance use, depression, anxiety, loneliness and others) at weeks 0, 8 (end of interveniton), 24 and 48. All participants in this arm will also receive a Fitbit to track objective activity (e.g. step counts).

This phase will pursue the following Aims:

Aim 1: Evaluate short (week 8) and longer term (weeks 12, 24) effectiveness of WE RISE on HIV (↑ ART adherence, ↑ continuous viral suppression), trauma (↓ trauma symptoms), substance use (↓ days and amount of substance use) and transdiagnostic factors such as mood (↓depression, ↓anxiety), stigma and loneliness.

Aim 2: Document the WE RISE implementation process by characterizing reach, effectiveness, adoption, implementation and maintenance (RE-AIM) by site for 24 weeks.

Phase 2 of WE RISE is an observational study that will focus on sustainability of WE RISE once research funding is completed. We will encourage our partnering community based organizations to adapt WE RISE as they see fit to enable them to continue to provide the intervention. Participants will undergo the same assessment schedule as in phase 1. In this phase, the study team will continue to observe and document the intervention for adaptations made and persistence of intervention fidelity.

This phase will focus on Aim 3.

Aim 3: Transcreate alternate or additional IS that address site specific barriers and facilitators to optimize the effectiveness, maintenance and broader dissemination of WE RISE at 24 weeks while documenting the implementation process (RE-AIM) and site-specific adaptations using the Framework for Recording Adaptations and Modifications-Enhanced (FRAME) through 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Is female sex at birth (cis-women)
2. Able to read and understand English
3. Able to participate in a low intensity exercise program
4. HIV-seropositive
5. At risk substance use (any illegal or unprescribed drug), tobacco, marijuana or alcohol use (four or more drinks in one day or 8 or more in one week).
6. Reports missing more ART doses than previous months, or > 5 in a month, or has a detectable HIV viral load
7. Experienced interpersonal violence
8. Able and willing to provide informed consent
9. Confirmed COVID-19 vaccinated x 2 or willingness to wear a mask during inperson interactions.

Exclusion Criteria:

1. Unwilling to participate in video record sessions (used to evaluate the quality of the intervention)
2. Enrolled in hospice
3. Not willing or not able to comply with study advisory board group participation agreement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Antiretroviral therapy (ART) adherence by drug levels | Weeks 0, 8, 24 and 48.
  All participants will undergo testing for ART in hair samples

SECONDARY OUTCOMES:
Antiretroviral therapy (ART) adherence by visual analog scale | Weeks 0, 8, 24 and 48.
  Self reported measure of adherence on a scale (score range 0 to 100 higher scores indicate higher adherence)
Generalized Anxiety Disorder-7 | Weeks 0, 8, 24 and 48.
  Measure of anxiety (score range 0 to 21, sum of items, 0-4 minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, 15-21 severe anxiety)
Patient Health Questionnaire - 9 | Weeks 0, 8, 24 and 48.
  Measure of depression (score range 0-27, sum of items, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression)
Timeline follow back substance use | Weekly during weeks 0-8, 24 and 48.
  Recall of substance use in the past week
International trauma questionnaire | Weeks 0, 8, 24 and 48.
  Provides two components of scoring and interpretation: 1) categorical scoring for the diagnosis of post traumatic stress disorder, PTSD (two or more question 1 or 2, two or more question 3 or 4, two of more question 5 or 6, two or more question 7,8,9) and complex post traumatic stress disorder, CPTSD (two or more question 10 or 11, two or more questions 12 or 13, two or more questions 14 or 15, two or more questions 16,17,18). 2) Dimensional scores from 0 to 24 (higher scores indicate higher symptom severity) are also presented for the two subscales. For PTSD sum items 1 to 6, for disturbances of self organization sum items 10 to 15.

OTHER OUTCOMES:
HIV Stigma Scale 12-short form | Weeks 0, 8, 24 and 48.
  Evaluates HIV stigma (scale ranges 12-48, sum of all items, higher scores indicate higher internalization of stigma)
Loneliness (UCLA-3 item) | Weeks 0, 8, 24 and 48.
  Three item question about loneliness (range 1-9, score is sum of all items, higher score indicates higher loneliness)
Fitbit data | Weeks 0, 8, 24 and 48.
  average step counts in past 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maile Karris, MD, Principal Investigator — UCSD
Locations (1):
- UC San Diego AntiViral Research Center (AVRC), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data (e.g. data alone without any possible identifying information) will be shared wit the NIMH data archive and the Sociostructural Implementation Science Coordination Initiative Hub for other researchers to access and use as per funding requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6-12 months of entry for the duration of the above mentioned databases.
Access Criteria: Access is dependent on the parent databases policy at the time of request.